CLINICAL TRIAL: NCT05200104
Title: An Open-label Phase 2a Study to Assess the Pharmacokinetics and Pharmacodynamic of PXL065 Parameters After 12 Weeks of Treatment in Male Subjects With Adrenomyeloneuropathy (AMN) Form of X-linked Adrenoleukodystrophy (X-ALD or ALD)
Brief Title: Study to Assess PXL065 in Subjects With Adrenomyeloneuropathy (AMN) Form of X-linked Adrenoleukodystrophy (X-ALD or ALD)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding unavailable
Sponsor: Poxel SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PXL065-005
Record Dates: First submitted 2022-01-06; First posted 2022-01-20 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: ALD (Adrenoleukodystrophy)
MeSH Terms: conditions — Adrenoleukodystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PXL065 (Experimental): PXL065 22.5 mg QD
  Interventions: Drug: PXL065

INTERVENTIONS:
Drug: PXL065 — PXL065 22.5 mg QD

SUMMARY:
A randomized open-label Phase 2a study to assess the pharmacokinetics and pharmacodynamic parameters of PXL065 after 12 weeks of treatment in male subjects with adrenomyeloneuropathy (AMN).

DETAILED DESCRIPTION:
A randomized open-label Phase 2a study to assess the pharmacokinetics and pharmacodynamic parameters of PXL065 after 12 weeks of treatment in male subjects with adrenomyeloneuropathy (AMN).

There will be a total of 3 study periods.

* Screening period of a maximum of 4 weeks prior to the open-label Treatment Period (Baseline Visit - V2). This period can be exceptionally extended for 2 weeks
* Open-label Treatment Period of 12 weeks
* Follow-up Period of 2 weeks after the last intake of the treatment (V5-End of Treatment Visit (EoT)).

During the treatment period, very long chain fatty acids (VLCFA) will be assessed every 4 weeks, to evaluate the kinetics of the PXL065 effect. Neurofilament light (NfL) will be assessed after 8 and 12 weeks of treatment, and other exploratory biomarkers after 12 weeks of treatment. A follow up period will allow continued monitoring the subjects' safety and evaluation of the kinetics of the 2 main biomarkers (VLCFA and NfL) at 2 weeks after the last intake of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with either a confirmed diagnosis of AMN by genetic testing (mutation in the ATP binding cassette subfamily D (ABCD1 gene)) or a family history of X-linked adrenoleukodystrophy (ALD) together with an elevation in VLCFA obtained from overnight fasting plasma sample at Screening Visit (V1).
* Age: ≥ 18 to ≤ 65 years at informed consent signature.
* Normal brain magnetic resonance imaging (MRI) or brain MRI showing non-specific abnormalities that can be observed in AMN subjects without signs of cerebral form of ALD (C-ALD). MRI must be performed within 6 months prior to V2. If there is no available brain MRI within this period, a brain MRI must be performed before V2

Exclusion Criteria:

* Any progressive neurological disease other than AMN.
* Arrested or progressing C-ALD as defined by cerebral lesions (except for non-specific abnormalities that can be observed in AMN subjects).
* Prior receipt of an allogeneic hematopoietic stem cell transplant or gene therapy

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic | Week 4
  Deuterated and protonated forms of (R)-pioglitazone and (S)-pioglitazone: Cmax
PharmacoKinetic | Week 4
  Deuterated and protonated forms of (R)-pioglitazone and (S)-pioglitazone: AUC0-24 (AUCtau)